CLINICAL TRIAL: NCT02042118
Title: Randomized Clinical Trial Assessing Laryngeal Mask Airway (LMA) Versus Face-mask Ventilation (FMV) in Neonatal Resuscitation at Mulago Hospital, Uganda
Brief Title: Randomized Clinical Trial Assessing Laryngeal Mask Airway Versus Face-mask Ventilation in Neonatal Resuscitation
Acronym: LMAvsFMV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre For International Health (Other)
Collaborators: Makerere University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LMAvsFMV
Record Dates: First submitted 2013-12-16; First posted 2014-01-22 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Asphyxia Neonatorum
Keywords: Neonatal resuscitation; Laryngeal Mask Airway (LMA); Face mask ventilation (FMV); Uganda; Africa
MeSH Terms: conditions — Asphyxia Neonatorum | interventions — Laryngeal Masks

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Laryngeal Mask Airway (Experimental): Laryngeal mask airway (LMA) ventilation will be provided for newborns in this arm during the first 2.5 minutes.
  Interventions: Device: Laryngeal Mask Airway
- Face mask ventilation (Active Comparator): Face-mask ventilation (FMV) will be provided for newborns in this arm during the first 2.5 minutes.
  Interventions: Device: Face mask ventilation

INTERVENTIONS:
Device: Laryngeal Mask Airway — Laryngeal mask airway (LMA) ventilation will be provided for newborns in this arm during the first 2.5 minutes.
  Other Names: I-gel size 1, Intersurgical Ltd, Wokingham, Berkshire,UK
  Arms: Laryngeal Mask Airway
Device: Face mask ventilation — Face-mask ventilation (FMV) will be provided for newborns in this arm during the first 2.5 minutes.
  Other Names: Face-mask ventilation; Neonatal resuscitator
  Arms: Face mask ventilation

SUMMARY:
The purpose of this study is to compare the use of a laryngeal mask airway (LMA) vs. face-mask ventilation (FMV) during first-line neonatal resuscitation in Mulago Hospital, Kampala, Uganda.

DETAILED DESCRIPTION:
Background: Perinatal mortality in Eastern Uganda 2007/2008 was estimated to 41/1000 pregnancies. The rate of stillbirth was 19/1000. In the whole of Uganda in 2008, neonatal deaths constituted 21% of an estimated 190,000 under five deaths, while HIV constituted only 5%. Implementing a Helping Babies Breathe (HBB) program in one centre in Tanzania resulted in almost 40 % reduction of early neonatal mortality. Introducing a neonatal intervention package even reduced the rate of stillbirths. Birth asphyxia (BA) accounted for 60% of early neonatal deaths in Haydom Lutheran Hospital, Tanzania.

The need for resuscitation is greater in the neonate than in any other age group. Providing effective positive pressure ventilation (PPV) is the single most important component of successful neonatal resuscitation (5). Ventilation is frequently initiated with face-mask ventilation (FMV) followed by endotracheal intubation (ETT) if depression continues. These techniques may be difficult to perform resulting in prolonged resuscitation. The laryngeal mask airway (LMA) may achieve initial ventilation and successful resuscitation faster than a face-mask device or ETT. Various publications and a Cochrane review has shown LMA to be as efficient as ETT. Important air leakage during FMV is an issue. LMA reduces the need for ETT. The latest generation of LMA is made of a medical-grade gel-like elastomer designed to provide an efficient seal to the larynx without an inflatable cuff. The risk for trauma is minimised. Insertion is easy with a low risk of tissue compression or dislodgement. In a study to evaluate educational intervention in the Democratic Republic of Congo, both physicians and midwifes showed a good level of expertise in LMA insertion on mannequins. Both groups almost unanimously manifested a high degree of approval of neonatal resuscitation with LMA.

Objective: To compare the use of uncuffed LMA vs. FMV during neonatal resuscitation in Mulago Hospital, Kampala, Uganda.

Study design, setting and population: A randomized clinical trial will be conducted in Mulago hospital among asphyxiated neonates in the delivery unit. Approximately 33000 babies are born in this hospital each year.

Prior to the intervention all staff in the labour ward performing resuscitation will receive training according to the HBB curriculum with a special module for training on LMA insertion.

A total of 50 neonates will be randomized into being resuscitated with FMV or LMA. A trained midwife under supervision of a paediatrician/anaesthesiologist will initiate the resuscitation. Data from the intervention will be recorded by a research assistant and by video. Resuscitation lasting more than 150 seconds will be handed over to the supervising physician. Resuscitation will be performed according to international guidelines.

Utility of study: Findings from this study will determine if uncuffed LMA can improve outcome of asphyxiated newborn in a large delivery ward where resuscitation is performed by midwifes. Data will also show us whether uncuffed LMA is superior to FMV after a training course according to the 2010 Guidelines on Neonatal Resuscitation (AHA, European Resuscitation Council [ERC], ILCOR). The Millennium Development Goals 4 (MDG-4) aims for the reduction of child mortality by two thirds from 1990 to 2015. It is crucial to explore alternative, cost-effective modalities that not only would reduce mortality, but also the burden of neurological damage in survivors.

ELIGIBILITY:
Inclusion Criteria:

* estimated gestation > 34 weeks
* estimated weight > 2000 gram
* need for Positive Pressure Ventilation (PPV) at birth

Exclusion Criteria:

* still birth
* major malformations
* severe prenatal depression (Heart rate <60 1 minute after birth)

Max Age: 1 Hour | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2015-05 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
time to spontaneous ventilation | one day
  To assess if the ventilation time needed for neonates with an estimated birth weight of 2 kg or above and in need of initial respiratory support can be decreased from an average of 132 seconds in infants being resuscitated using FMV (control arm) to an average ventilation time of 72 seconds for infants resuscitated with the use of LMA (interventions arm).

SECONDARY OUTCOMES:
proportion of infants who require advanced resuscitation | 1 day
  To determine if use of LMA can reduce the proportion of infants who require advanced resuscitation
the proportion of infants with adverse birth outcome | 2 days
  To assess the proportion of infants with adverse outcome (death or hospitalization) at 24 and 48 hours of life.

OTHER OUTCOMES:
Proportion of times the midwife successfully inserts the LMA and deliver efficient PPV | 1 day
  To determine if midwifes can learn to insert LMA and deliver efficient PPV.
Proportion of times the midwife successfully deliver efficient PPV using FMV | 1 day
  To determine the best way for midwifes that have gone through the Helping Babies Breathe (HBB) curriculum to deliver PPV
proportion of video recordings that provides the necessary elements for QA | 1 day
  To determine if video recording can be used for Quality assurance (QA) of resuscitation and data collection.

CONTACTS AND LOCATIONS:
Overall Officials: Thorkild Tylleskar, MD, PhD, Study Chair — Centre for International Health, University of Bergen; Nicolas J Pejovic, MD, Principal Investigator — Centre for International Health, University of Bergen
Locations (1):
- Mulago Teaching Hospital, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ersdal HL, Mduma E, Svensen E, Perlman J. Birth asphyxia: a major cause of early neonatal mortality in a Tanzanian rural hospital. Pediatrics. 2012 May;129(5):e1238-43. doi: 10.1542/peds.2011-3134. Epub 2012 Apr 16. PMID 22508912
- [Background] Ersdal HL, Mduma E, Svensen E, Perlman JM. Early initiation of basic resuscitation interventions including face mask ventilation may reduce birth asphyxia related mortality in low-income countries: a prospective descriptive observational study. Resuscitation. 2012 Jul;83(7):869-73. doi: 10.1016/j.resuscitation.2011.12.011. Epub 2011 Dec 23. PMID 22198423
- [Background] Grein AJ, Weiner GM. Laryngeal mask airway versus bag-mask ventilation or endotracheal intubation for neonatal resuscitation. Cochrane Database Syst Rev. 2005 Apr 18;(2):CD003314. doi: 10.1002/14651858.CD003314.pub2. PMID 15846656
- [Background] Zhu XY, Lin BC, Zhang QS, Ye HM, Yu RJ. A prospective evaluation of the efficacy of the laryngeal mask airway during neonatal resuscitation. Resuscitation. 2011 Nov;82(11):1405-9. doi: 10.1016/j.resuscitation.2011.06.010. Epub 2011 Jul 16. PMID 21763393
- [Background] Carbine DN, Finer NN, Knodel E, Rich W. Video recording as a means of evaluating neonatal resuscitation performance. Pediatrics. 2000 Oct;106(4):654-8. doi: 10.1542/peds.106.4.654. PMID 11015505
- [Background] Nankabirwa V, Tumwine JK, Tylleskar T, Nankunda J, Sommerfelt H; PROMISE EBF Research Consortium. Perinatal mortality in eastern Uganda: a community based prospective cohort study. PLoS One. 2011 May 9;6(5):e19674. doi: 10.1371/journal.pone.0019674. PMID 21573019
- [Result] Pejovic NJ, Trevisanuto D, Nankunda J, Tylleskar T. Pilot manikin study showed that a supraglottic airway device improved simulated neonatal ventilation in a low-resource setting. Acta Paediatr. 2016 Dec;105(12):1440-1443. doi: 10.1111/apa.13565. PMID 27582031
- [Derived] Pejovic NJ, Trevisanuto D, Lubulwa C, Myrnerts Hook S, Cavallin F, Byamugisha J, Nankunda J, Tylleskar T. Neonatal resuscitation using a laryngeal mask airway: a randomised trial in Uganda. Arch Dis Child. 2018 Mar;103(3):255-260. doi: 10.1136/archdischild-2017-312934. Epub 2017 Sep 14. PMID 28912163